CLINICAL TRIAL: NCT01483456
Title: A Multidisciplinary Program for Preventing Falls "Identify, Prevent and Get up": Impact on Falls in Elderly Inpatients
Brief Title: Impact of Multidisciplinary Program on Falls in Elderly Inpatients
Acronym: IPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011.666
Record Dates: First submitted 2011-07-21; First posted 2011-12-01 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Falls Among Elderly Inpatients
Keywords: Accidental falls; safety management; aged; inpatient; stepped wedge design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual care (Other)
  Interventions: Other: The multidisciplinary prevention program called "IPR" (in French "Identifier, Prévenir, Relever")

INTERVENTIONS:
Other: The multidisciplinary prevention program called "IPR" (in French "Identifier, Prévenir, Relever") — The intervention is a multidisciplinary program of fall prevention including 3 complementary interventions which focus on several stages of elderly inpatient management:
  1. Identification of patient's fall risk,
  2. Multifactorial fall prevention program (integrated actions targeted on risk factors, exercise programs and review of the hospital environment),
  3. "Get up" workshop and morbidity and mortality conferences related to fall cases

SUMMARY:
Falls among elderly inpatients are common, multifactorial and associated with a significant increase of complications and morbidity. According to a recent Cochrane review, the effectiveness of fall prevention program has been assessed in community-dwelling and in long stay wards but not in rehabilitation wards (RW) and geriatric acute wards (GAW). IPR study aims to measure the impact of a multidisciplinary prevention program on falls in elderly inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged over 65 years
* Admitted during the study
* Participation agreement

Exclusion Criteria:

* Patients with a MMSE<10 and incapable to participate to a reeducation program
* Patient with an evolutionary and\or badly checked psychiatric pathology
* Bedridden patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1852 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of falls among elderly inpatients | patients will be followed for the duration of hospital stay, 15 months maximum

SECONDARY OUTCOMES:
Incidence of fall-related mortality | patients will be followed for the duration of hospital stay, 15 months maximum
Incidence of fall-related | patients will be followed for the duration of hospital stay, 15 months maximum

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KROLAK-SALMON, Principal Investigator — Hospices Civils de Lyon
Locations (12):
- France (12):
  - Centre Hospitalier Gériatrique du Mont d'Or, Albigny-sur-Saône
  - Centre Hospitalier d'Ardèche Méridionale - Service de Gériatrie, Centre Hospitalier d'Ardèche Méridionale, Aubenas
  - Centre Hospitalier de Bourg en Bresse - Pôle filière gériatrique, Centre Hospitalier de Bourg en Bresse, Bourg-en-Bresse
  - Hospices Civils de Lyon - Hôpital Frédérique Dugoujon, Caluire-et-Cuire
  - Hospices Civils de Lyon - Hôpital Antoine Charial, Francheville
  - Hospices Civils de Lyon - Hôpital Pierre Garraud, Lyon
  - Hospices Civils de Lyon - Service de Médecine gériatrique, Hôpital Edouard Herriot, Lyon
  - Hôpital Local de Meximieux, Meximieux
  - Hospices Civils de Lyon - Service de Médecine gériatrique, Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier d'Annecy - Pôle de Gériatrie - Centre Hospitalier d'Annecy, Pringy
  - Centre Hospitalier Lucien Hussel - Pôle gérontologie, Vienne
  - Hospices Civils de Lyon - Service de Gériatrie - Hôpital des Charpennes, Villeurbanne